CLINICAL TRIAL: NCT02330926
Title: A Randomised, Open-label Trial of a Multimodal Intervention (Exercise, Nutrition and Antiinflammatory Medication) Plus Standard Care Versus Standard Care Alone to Prevent/Attenuate Cachexia in Advanced Cancer Patients Undergoing Chemotherapy
Brief Title: Multimodal Intervention for Cachexia in Advanced Cancer Patients Undergoing Chemotherapy
Acronym: MENAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Oslo University Hospital (Other); Cantonal Hospital of St. Gallen (Other); Ottawa Regional Cancer Centre (Other); Jewish General Hospital (Other); Cross Cancer Institute (Other); The Beatson West of Scotland Cancer Centre (Unknown); Queen Margaret Hospital, Dunfermline (Other); Cancer Research UK Edinburgh Centre (Unknown); Malteser Krankenhaus Seliger Gerhardt (Unknown); Tumor Biology Center Freiburg (Unknown); Tumor Zentrum Aarau (Unknown); Chelsea and Westminster NHS Foundation Trust (Other); Cedars-Sinai Medical Center (Other); Guy's and St Thomas' NHS Foundation Trust (Other); NHS Forth Valley (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MENAC-2013-05; 2013-002282-19 (EudraCT Number)
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cachexia; Neoplasms
Keywords: Combined modality treatment; Diet therapy; Exercise therapy; Ibuprofen; Dietary supplements
MeSH Terms: conditions — Cachexia; Neoplasms | interventions — Standard of Care; Dietary Supplements; Counseling; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- multimodal intervention (Experimental): standard care plus multimodal intervention consisting of nutritional supplements and advice, home-based self-assisted exercise program, and anti-inflammatory medication (ibuprofen)
  Interventions: Other: standard care; Dietary Supplement: nutritional supplements and advice; Behavioral: home-based self-assisted exercise program; Drug: Ibuprofen
- standard care (Active Comparator): standard palliative care
  Interventions: Other: standard care

INTERVENTIONS:
Other: standard care — Routine oncology and palliative care
Dietary Supplement: nutritional supplements and advice — n-3 PUFA enriched supplements, dietary advice
  Arms: multimodal intervention
Behavioral: home-based self-assisted exercise program — Strength and aerobic
  Arms: multimodal intervention
Drug: Ibuprofen — 400mgx3
  Arms: multimodal intervention

SUMMARY:
Cancer cachexia is a multi-factorial syndrome defined by an ongoing loss of skeletal muscle mass (with or without loss of fat mass) that cannot be fully reversed by conventional nutritional support and leads to progressive functional impairment.

There is an urgency for improving management, but there is no consensus on the optimal treatment for cancer cachexia. Several single therapies for cancer cachexia have been examined in clinical trials, with disappointing overall results. As multiple factors are responsible for the development of cachexia, it has been argued that optimal cachexia interventions should target all components: multimodal therapy for a multimodal problem.

The overall aim of this study is to early prevent the development of cachexia rather than treatment late in the disease trajectory. From a patient perspective a short term effect will be to improve physical and psychological function, to reduce symptom burden and to improve survival. In other words live a longer and better life during and after chemotherapy. Direct effects of the cachexia intervention are expected to be reduction of weight and muscle loss, and improved physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lung cancer, pancreatic cancer or cholangiocarcinoma where the diagnosis is based on histological, radiological or multidisciplinary team (MDT) evaluation
* non-small cell lung cancer (stage III or IV), pancreatic adenocarcinoma (stage III or IV), due to commence first or second line anticancer treatment (defined as chemotherapy, chemo-radiotherapy, targeted therapy or immunotherapy)
* staging CT within 4 weeks of commencement of anti-cancer therapy (in patients where staging CT is out-with this period, further CT scanning will be undertaken. PETCT's are also appropriate)
* completed all other baseline assessments within one week prior to first course of anti-cancer treatment
* written informed consent
* able to comply with trial interventions (in the opinion of referring clinician) e.g. willing and able to do light exercise and take oral nutritional supplements as well as no major contraindications against ibuprofen.
* Karnofsky Performance Status >70

Exclusion Criteria:

* Neuro-endocrine pancreatic cancer
* Creatinine clearance <30ml/min
* Receiving parenteral nutrition or enteral nutrition via feeding tube
* receiving neo-adjuvant anti-cancer therapy
* BMI >30 kg/m2
* Use of appetite stimulants or anabolic/anti-catabolic agents (such as megestrol acetate, progestational agents, marijuana growth hormone, dronabinol, or other anabolic agent) within 30 days prior to study baseline
* Concomitant steroid (>10mg/d prednisolone or equivalent) treatment for less than three months prior to inclusion (inhaled, optical or pulsed oral steroids (up to 10 days use) are permitted)
* Concomitant long term (>1 week) nonsteroidal anti-inflammatory drugs (NSAID) or aspirin treatment
* pregnancy, breast-feeding or of child bearing potential (that is not postmenopausal or permanently sterilised) age and not using adequate contraception (oral, injected, implanted or hormonal methods of contraception, intrauterine device and barrier method)
* Concomitant anti-coagulant treatment (e.g. warfarin or heparin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
change in body weight | 6 weeks
  body weight (Kg)

SECONDARY OUTCOMES:
change in muscle mass | 6 weeks
  CT L3 cross sectional area
change in physical activity | 6 weeks
  ActivPAL step count

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD PhD, Study Director — European Palliative Care Research Centre (PRC), Department of Cancer Research and Molecular Medicine, Faculty of Medicine, NTNU, Trondheim, Norway; Marie Fallon, MD PhD, Study Director — Edinburgh Cancer Research Centre, University of Edinburgh, Edinburgh, UK
Locations (17):
- Cedars-Sinai Medical Center, Los Angeles, California, United States
- Canada (4):
  - CA4 Brampton Civic Hospital, Brampton
  - Cross Cancer Insitute, Edmonton
  - Jewish General Hospital, Montreal
  - Ottawa Regional Cancer Centre, Ottawa
- Universitätsklinikum Bonn, Bonn, Germany
- Norway (2):
  - Oslo University Hospital, Oslo
  - St Olavs Hospital, Trondheim
- Switzerland (2):
  - Tumor Zentrum, Aarau
  - Cantonal Hospital, Sankt Gallen
- United Kingdom (7):
  - NHS Forth Valley, Larbert, Falkirk
  - Queen Margaret Hospital, Dunfermline, Fife
  - Llandough Hospital, Cardiff
  - Edinburgh Cancer Centre, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Chelsea and Westminister Hospital NHS, London
  - Guys and St Thomas, London

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Solheim TS, Laird BJA, Balstad TR, Bye A, Stene G, Baracos V, Strasser F, Griffiths G, Maddocks M, Fallon M, Kaasa S, Fearon K. Cancer cachexia: rationale for the MENAC (Multimodal-Exercise, Nutrition and Anti-inflammatory medication for Cachexia) trial. BMJ Support Palliat Care. 2018 Sep;8(3):258-265. doi: 10.1136/bmjspcare-2017-001440. Epub 2018 Feb 9. PMID 29440149
- [Derived] Naito T. Challenges in enhancing physical performance in thoracic cancer cachexia. Thorac Cancer. 2021 Oct;12(20):2633-2634. doi: 10.1111/1759-7714.14154. Epub 2021 Sep 15. No abstract available. PMID 34528401

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT02330926/SAP_000.pdf